CLINICAL TRIAL: NCT01811381
Title: Curcumin and Yoga Exercise Effects in Veterans at Risk for Alzheimer's Disease
Brief Title: Curcumin and Yoga Therapy for Those at Risk for Alzheimer's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: E0669-I; VA_RX00069 (Other Grant/Funding Number: Veterans Affairs)
Record Dates: First submitted 2013-02-11; First posted 2013-03-14 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Mild Cognitive Impairment
Keywords: Alzheimer; Prevention; mild cognitive impairment; physical exercise; synergism; curcumin; dietary supplement; anti-inflammatory; anti-tau; subjective memory complaints without MCI; plasma-exosomes; plasm- extracellular-derived-vesicles
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Curcumin and aerobic exercise (Experimental): For the first 6 months of the study, subjects will take 800 mg of curcumin (4 capsules x BID, p.o.) before meals. From six to 12 months after the beginning of the study, subjects will take curcumin (4 capsules BID before meals, total 800 mg/day) and also participate in an aerobic yoga exercise program (Attendance at 2 classes of 1 hour duration [or 1 hr SecureVideo Live videoconference remote classes for subject who become proficient] and 2 home practices of 30 minute duration per week).
  Interventions: Drug: Curcumin; Behavioral: aerobic yoga
- Placebo vs non-aerobic yoga (Placebo Comparator): For the first 6 months of the study, subjects will take Placebo (4 capsules x BID, p.o.) before meals. From six months to 12 months from the beginning of the study, subjects will take Placebo (4 capsules x BID) and participate in a weekly non-aerobic yoga program (Attendance at 2 classes of 1 hour duration or 1 hr SecureVideo Live videoconference remote classes for subject who become proficient] and 2 home practices of 30 minute duration per week).
  Interventions: Behavioral: non aerobic yoga; Dietary Supplement: Placebo
- Placebo vs Aerobic Yoga (Active Comparator): For the first 6 months of the study, subjects will take Placebo (4 capsules x BID, p.o.) before meals. From six months to 12 months from the beginning of the study, subjects will take Placebo (4 capsules x BID) and participate in a weekly aerobic yoga program (Attendance at 2 classes of 1 hour duration [or 1 hr SecureVideo Live videoconference remote classes for subject who become proficient] and 2 home practices of 30 minute duration per week).
  Interventions: Behavioral: aerobic yoga; Dietary Supplement: Placebo
- Curcumin vs non aerobic yoga (Active Comparator): For the first 6 months of the study, subjects will take 800 mg of curcumin (4 capsules x BID, p.o.) before meals. From six months to 12 months from the beginning of the study, subjects will take Curcumin (4 capsules x BID, total 800 mg/day) and participate in a weekly non-aerobic yoga program (Attendance at 2 classes of 1 hour duration [or 1 hr SecureVideo Live videoconference remote classes for subject who become proficient] and 2 home practices of 30 minute duration per week).
  Interventions: Drug: Curcumin; Behavioral: aerobic yoga

INTERVENTIONS:
Drug: Curcumin — Subjects will take 800 mg of curcumin in 4 capsules BID per day prior to meals
  Other Names: Longvida Curcumin (Verdure Sciences, Indianapolis)
  Arms: Curcumin and aerobic exercise; Curcumin vs non aerobic yoga
Behavioral: aerobic yoga — Each week, subjects will attend two one hour aerobic yoga classes under the supervision of certified yoga instructors and complete two 30 minute aerobic yoga practice sessions at home. If proficient, subjects will take a live-video conference remote class, HIPAA approved SecureVideo classes. Modification of consent has been approved.
  Arms: Curcumin and aerobic exercise; Curcumin vs non aerobic yoga; Placebo vs Aerobic Yoga
Behavioral: non aerobic yoga — Subjects will take two non-aerobic (stretching) classes weekly as well as practice two 30 minutes yoga routines at home weekly.
  Each week, subjects will attend two one hour non-aerobic yoga classes under the supervision of certified yoga instructors and complete two 30 minute non-aerobic yoga practice sessions at home.
  Arms: Placebo vs non-aerobic yoga
Dietary Supplement: Placebo — Subjects will take 4 capsules x BID of placebo
  Arms: Placebo vs Aerobic Yoga; Placebo vs non-aerobic yoga

SUMMARY:
Physical exercise has proven to improve memory including in the elderly. Drugs developed to stop the underlying disease processes that cause Alzheimer's disease may succeed only with multimodal efforts to stimulate brain function. One purpose of the study is to test the clinical benefits of curcumin, a safe and effective compound isolated from the turmeric root (a component of Indian curry spices), which has been found to inhibit several potential disease pathways in Alzheimer's disease. Another purpose of this study is to determine how the addition of a physical exercise program in individuals with early memory problems may affect memory function or brain imaging and blood-based markers associated with Alzheimer's disease.

DETAILED DESCRIPTION:
Subjects with Mild cognitive impairment (MCI) or Subjective Cognitive Impairment (SCD) are eligible for this study. MCI often represents the earliest stages of Alzheimer's disease (AD), as individuals meeting criteria for MCI are subsequently diagnosed with AD at much higher rates than their cognitively normal elderly peers. Subjects with MCI are at risk of developing AD, within 6 years. Subjects with SCD may be at risk to develop MCI. The study is stratified according to whether subjects have SCD or MCI. The goal of the current study is to determine whether dietary supplementation with a novel formulation of curcumin (a component of the curry spice turmeric), which is better absorbed and more efficiently transported into the brain, can alter biological and clinical markers associated with AD risk, and to determine whether the potential beneficial effects of curcumin supplementation are synergistic with aerobic exercise. The investigators will recruit 80 elderly participants meeting criteria for MCI. Over the second 6 months of the study, the curcumin and placebo groups will be further divided into groups receiving training in either aerobic or non-aerobic yoga to determine the synergism between curcumin supplementation and aerobic exercise. The effectiveness of these interventions will be measured using plasma samples (for expression of Alzheimer-related biomarkers), and neuropsychological, functional, and behavioral assessments (i.e. clinical measures) collected at baseline, 6 months, and 12 months after initiation of treatments, with a subset of participants receiving brain imaging at baseline and 6 months. Dosage is titered up two weeks prior to study start (1 capsule BID, first five days, then 2 capsules BID for five days, then 6 capsules BID for five days, then 8 capsules BID- study dosage). Over the first 6 months of the study, participants will be randomized into equal groups receiving dietary supplementation with either curcumin or placebo. Patients are stratified according to whether they have only subjective memory complaints without MCI versus those that have MCI. Over the second 6 months of the study, participants will be further randomized into equal groups receiving dietary supplementation with either curcumin or placebo.

ELIGIBILITY:
Inclusion Criteria:

* age between 50 and 90 years;
* Mini-Mental Status Exam (MMSE) scores greater than 24;
* subjective cognitive complaints based on subjective cognitive impairment questionaire (Gifford et al. 2015) including non-amnestic or amnestic cognitive deficits MCI (performance 1.5 standard deviation (SD) below normative means on The Consortium to Establish a Registry for Alzheimer's Disease (CERAD) word list learning test);
* essentially intact activities of daily living (FAQ scores < 6);
* Sedentary (exercise < 30 minutes a day, 3 times a week);
* ambulatory, able exercise safely without cardiovascular symptoms, and able to pass a graded treadmill test modified for the elderly;
* able to arrange transportation to the study;
* Willing and intellectually able to understand and to sign an informed consent and to adhere to protocol requirements;
* community dwelling; and
* fluent in written and spoken English
* must screen positive for a Modified abbreviated MCI or SCD screen on phone, before coming in to clinic for extensive testing

Exclusion Criteria:

* diagnosis of dementia,
* concurrent substance abuse disorder,
* psychosis or mood disorder,
* neurological disease affecting motor or cognitive abilities (e.g. Parkinson's disease),or other significant uncontrolled medical problems,
* cannot get up and down from floor
* initiation of any new medications/treatment for cognitive impairment (i.e. cholinesterase inhibitor, memantine) < 6 months prior to study enrollment

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female subjects have the same inclusion and exclusion criteria as men. Although males have increased representation in the veteran population, which is prioritized, we make efforts to recruit females through the LA times.
Enrollment: 80 (Estimated)
Dates: Start 2014-01-20 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Curcumin effects (first six month period) or curcumin and aerobic yoga effects (second six month period) on the changes in the levels of blood biomarkers for Mild Cognitive Impairment relative to baseline or relative to placebo or non-aerobic yoga. | 0, 6, and 12 months
  Blood samples at baseline & follow-ups are collected & analyzed for changes in biomarkers associated with MCI and/or curcumin: Clusterin, C-reactive protein, N-terminal prohormone of brain natriuretic peptide, Apolipoprotein E, beta-amyloid, vascular cell adhesion molecule protein-1, Brain derived neurotrophic factor, Interleukin-6, Interleukin-1 beta, Interleukin 1 receptor accessory protein-like 2, Tumor necrosis factor alpha, Osteopontin. The investigators will test whether supplements and/or exercise type are associated with a decrease in the biomarkers thought to be associated with MCI

SECONDARY OUTCOMES:
Changes in 18F-fluorodeoxyglucose (FDG) Positron Emission Tomography (PET) glucose metabolism neuroimaging after supplementation compared to baseline and compared to placebo | 0 and 6 months
  Functional connectivity multivariate discriminant analysis of neuroimaging changes using 18FDG-PET predicting rapid conversion to Alzheimer will be examined in subjects on supplements compared to those on placebo. Cerebral metabolism of glucose will be assessed for those receiving supplements vs. placebo and vs baseline (first six months).
Curcumin effects on changes in Neuropsychological parameters compared to baseline and to placebo (first six month period) and in combination with aerobic yoga, compared to baseline and to non-aerobic yoga with curcumin or aerobic yoga with supplement | 0, 6, 12 months
  Cognitive changes shown to precede Alzheimer's will be assessed using a neuropsychological battery. Behavioral symptoms will be assessed with the Neuropsychiatric Inventory Questionnaire (NPI-Q). Instrumental activities of daily living will be assessed with the Functional Activities Questionnaire. Overall assessment of disease severity will be assessed with the Clinical Dementia Rating Scale Sum of Boxes. subjects on supplements compared to those on placebo. Neuropsychiatric parameters will be assessed for those receiving supplements vs baseline or vs placebo or with those performing aerobic yoga with placebo or non aerobic yoga with curcumin (second six month period).
Number of Participants with Adverse Events | 0,3,6,9,12 months
  The investigators will perform routine comprehensive blood panel test to monitor safety and tolerability of Curcumin in subjects at risk for MCI by means of adverse events, vital signs and safety laboratory assessments. [ Time Frame: is at each timepoint in the study, 3, 6, 9 and 12 months].

CONTACTS AND LOCATIONS:
Overall Officials: Sally A Frautschy, PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: January 1, 2020 is our deadline to published the data.
Access Criteria: we will share data in a publication (biomarker data, curcumin pharmacokinetics, cognitive and neuroimaging changes). we may also provide RNAseq data on exosomes.

REFERENCES:
- [Background] Begum AN, Jones MR, Lim GP, Morihara T, Kim P, Heath DD, Rock CL, Pruitt MA, Yang F, Hudspeth B, Hu S, Faull KF, Teter B, Cole GM, Frautschy SA. Curcumin structure-function, bioavailability, and efficacy in models of neuroinflammation and Alzheimer's disease. J Pharmacol Exp Ther. 2008 Jul;326(1):196-208. doi: 10.1124/jpet.108.137455. Epub 2008 Apr 16. PMID 18417733
- [Background] Frautschy SA, Cole GM. Why pleiotropic interventions are needed for Alzheimer's disease. Mol Neurobiol. 2010 Jun;41(2-3):392-409. doi: 10.1007/s12035-010-8137-1. Epub 2010 May 2. PMID 20437209
- [Background] Frautschy SA, Hu W, Kim P, Miller SA, Chu T, Harris-White ME, Cole GM. Phenolic anti-inflammatory antioxidant reversal of Abeta-induced cognitive deficits and neuropathology. Neurobiol Aging. 2001 Nov-Dec;22(6):993-1005. doi: 10.1016/s0197-4580(01)00300-1. PMID 11755008
- [Background] Garcia-Alloza M, Borrelli LA, Rozkalne A, Hyman BT, Bacskai BJ. Curcumin labels amyloid pathology in vivo, disrupts existing plaques, and partially restores distorted neurites in an Alzheimer mouse model. J Neurochem. 2007 Aug;102(4):1095-104. doi: 10.1111/j.1471-4159.2007.04613.x. Epub 2007 Apr 30. PMID 17472706
- [Background] Geda YE, Roberts RO, Knopman DS, Christianson TJ, Pankratz VS, Ivnik RJ, Boeve BF, Tangalos EG, Petersen RC, Rocca WA. Physical exercise, aging, and mild cognitive impairment: a population-based study. Arch Neurol. 2010 Jan;67(1):80-6. doi: 10.1001/archneurol.2009.297. PMID 20065133
- [Background] Gota VS, Maru GB, Soni TG, Gandhi TR, Kochar N, Agarwal MG. Safety and pharmacokinetics of a solid lipid curcumin particle formulation in osteosarcoma patients and healthy volunteers. J Agric Food Chem. 2010 Feb 24;58(4):2095-9. doi: 10.1021/jf9024807. PMID 20092313
- [Background] Jankowsky JL, Melnikova T, Fadale DJ, Xu GM, Slunt HH, Gonzales V, Younkin LH, Younkin SG, Borchelt DR, Savonenko AV. Environmental enrichment mitigates cognitive deficits in a mouse model of Alzheimer's disease. J Neurosci. 2005 May 25;25(21):5217-24. doi: 10.1523/JNEUROSCI.5080-04.2005. PMID 15917461
- [Background] Lazarov O, Robinson J, Tang YP, Hairston IS, Korade-Mirnics Z, Lee VM, Hersh LB, Sapolsky RM, Mirnics K, Sisodia SS. Environmental enrichment reduces Abeta levels and amyloid deposition in transgenic mice. Cell. 2005 Mar 11;120(5):701-13. doi: 10.1016/j.cell.2005.01.015. PMID 15766532
- [Background] Liang KY, Mintun MA, Fagan AM, Goate AM, Bugg JM, Holtzman DM, Morris JC, Head D. Exercise and Alzheimer's disease biomarkers in cognitively normal older adults. Ann Neurol. 2010 Sep;68(3):311-8. doi: 10.1002/ana.22096. PMID 20818789
- [Background] Lim GP, Chu T, Yang F, Beech W, Frautschy SA, Cole GM. The curry spice curcumin reduces oxidative damage and amyloid pathology in an Alzheimer transgenic mouse. J Neurosci. 2001 Nov 1;21(21):8370-7. doi: 10.1523/JNEUROSCI.21-21-08370.2001. PMID 11606625
- [Background] Ma QL, Yang F, Rosario ER, Ubeda OJ, Beech W, Gant DJ, Chen PP, Hudspeth B, Chen C, Zhao Y, Vinters HV, Frautschy SA, Cole GM. Beta-amyloid oligomers induce phosphorylation of tau and inactivation of insulin receptor substrate via c-Jun N-terminal kinase signaling: suppression by omega-3 fatty acids and curcumin. J Neurosci. 2009 Jul 15;29(28):9078-89. doi: 10.1523/JNEUROSCI.1071-09.2009. PMID 19605645
- [Background] Scarmeas N, Luchsinger JA, Brickman AM, Cosentino S, Schupf N, Xin-Tang M, Gu Y, Stern Y. Physical activity and Alzheimer disease course. Am J Geriatr Psychiatry. 2011 May;19(5):471-81. doi: 10.1097/JGP.0b013e3181eb00a9. PMID 20808142
- [Background] Yang F, Lim GP, Begum AN, Ubeda OJ, Simmons MR, Ambegaokar SS, Chen PP, Kayed R, Glabe CG, Frautschy SA, Cole GM. Curcumin inhibits formation of amyloid beta oligomers and fibrils, binds plaques, and reduces amyloid in vivo. J Biol Chem. 2005 Feb 18;280(7):5892-901. doi: 10.1074/jbc.M404751200. Epub 2004 Dec 7. PMID 15590663
- [Background] Gifford KA, Liu D, Romano R 3rd, Jones RN, Jefferson AL. Development of a subjective cognitive decline questionnaire using item response theory: a pilot study. Alzheimers Dement (Amst). 2015 Dec 1;1(4):429-439. doi: 10.1016/j.dadm.2015.09.004. PMID 26878034
- See also: Improving care of Veterans — http://www.research.va.gov/